CLINICAL TRIAL: NCT03542708
Title: Prospectively Randomized Study of Intraovarian Injections of Autologous Platelet-rich Plasma (PRP) in Women With Primary Ovarian Insufficiency (POI)
Brief Title: Injections of Autologous PRP in Women With Primary Ovarian Insufficiency
Acronym: PRP4POI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Human Reproduction (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03192018-01
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-04

CONDITIONS: Primary Ovarian Insufficiency; Premature Menopause
MeSH Terms: conditions — Primary Ovarian Insufficiency; Menopause, Premature

STUDY DESIGN:
Intervention Model Description: One ovary will be randomly selected for treatment with PRP. The other ovary will serve as a control.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The care provider will be aware of which ovary is being treated. A different physician will serve as the outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-PRP (Experimental): The cortex of selected ovary will be injected with autologous platelet rich plasma.
  Interventions: Procedure: A-PRP
- Control (No Intervention): The contralateral ovary will not be injected.

INTERVENTIONS:
Procedure: A-PRP — The cortex of selected ovary will be injected with autologous platelet rich plasma. Up to ten different sites will be injected under ultrasound guidance. The patient will be under IV sedation. Record of which ovary was injected will be kept in the online research database and not in the clinical chart.
  Other Names: Autologous Platelet Rich Plasma
  Arms: A-PRP

SUMMARY:
Premature ovarian failure is a loss of normal function before age 40, leading to infertility and hypoestrogenism. This study will involve only adult women with a diagnosis of POI. Participants will receive injections of autologous PRP in one randomly selected ovary.

DETAILED DESCRIPTION:
Premature ovarian failure is a loss of normal function before age 40, leading to infertility and hypoestrogenism. While POI is sometimes called premature menopause, it is not the same thing as menopause. Women with POI may still have occasional irregular periods and may even occasionally achieve a pregnancy. Symptoms of POI include: irregular menses or amenorrhea, infertility, hypoestrogenic symptoms and decreased libido. POI may be caused by Chromosomal defects such as mosaic Turner's syndrome, exposure to toxins (chemotherapy or radiation), autoimmunity, genetic factors (FMR1) and other unknown factors.

Autologous Platelet Rich Plasma (A-PRP) is plasma with a concentration of platelets above the blood baseline. A-PRP is developed from autologous blood. Within A-PRP, the concentration of platelets delivers an increased number of growth factors. In this study A-PRP will be prepared using Regen Lab PRP Kit which is approved by US-FDA for preparation of PRP.

PRP is becoming widely used in a variety of medical procedures seeking tissue remodeling and/or healing as an intervention. To date, applications in orthopedics, wound healing, dermatology and plastic surgery have gained general acceptance, primarily as the role of platelets and their activation in tissue repair and recovery has become better understood at a cellular and molecular level. This knowledge base provides a foundation for the present study because of the ready availability of FDA-approved kits for autologous PRP preparations and the recognition that the aging ovary acquires tissue pathologies in the form of wound healing and fibrosis as a result of repeat ovulations over the reproductive lifespan of women. Since PRP is an autologous blood product, and is widely used via injection into various organs and tissues, safety concerns are minimal.

This study will involve only adult women with a diagnosis of POI. Consenting participants will receive injections of autologous Platelet RIch Plasma (A-PRP) in one randomly selected ovary under ultrasound guidance performed after induction of IV sedation. Randomization will determine whether the right or left ovary will be treated. The result of randomization will not be recorded in the participants clinical chart, but will be maintained in the research database with blinding to all clinical participants. The physician performing the A-PRP administration will not perform post procedure follow-up of those patients. In case of a complication, possibly related to treatment, the case will be unblinded.

The study will be powered to detect a 20% response in the treated ovary (every patient's 2nd ovary will serve as control). This will require 68 ovaries and 34 patients. The study, thus, does not involve randomization of patients because each patient's second ovary functions as control ovary, although which ovary will receive treatment in a given patient will be determined by computer randomization.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Women 40 years of age and younger with documented primary ovarian insufficiency.
* Normal Karyotype
* FSH > 30
* AMH not detectable
* No evidence of follicles > 4mm
* Must have two ovaries of approximately equal volume.
* No Aspirin or any NSAID (e.g. Motrin) for approximately one week before treatment
* Willingness to undergo further fertility treatment, including IVF if there is evidence of response

Exclusion Criteria:

* Premature ovarian failure due to a genetic origin, such as Turner's Syndrome or chromosomal abnormality
* Marked thrombocytopenia
* Blood diseases
* Hypofibrinogenemia
* Hemodynamic instability
* Anticoagulant or antiaggregant treatment
* Oncological diseases (specially, skeletal system and blood)
* Sepsis
* Acute and chronic infectious diseases
* Autoimmune diseases, for example, lupus erythematosus, etc.
* Active substance abuse or dependence
* Major Mental health disorder

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Ovarian Follicles | Change from baseline to 12 weeks
  Emergence of new ovarian follicles with evidence of estradiol production

SECONDARY OUTCOMES:
Increase in serum AMH | Change from baseline to 12 weeks
  Increase in serum AMH above baseline level
Retrieval of oocytes in an IVF cycle | 6 months
  Retrieval of oocytes in an IVF cycle
Clinical Pregnancy | 12 months
  Establishment of a Clinical pregnancy,

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Gleicher, MD, Principal Investigator — Medical Director
Locations (1):
- Center For Human Reproduction, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).